CLINICAL TRIAL: NCT01193088
Title: Genetics of Charcot Marie Tooth Disease (CMT) - Modifiers of CMT1A, New Causes of CMT
Brief Title: Genetics of Charcot Marie Tooth (CMT) - Modifiers of CMT1A, New Causes of CMT2
Acronym: INC-6602
Status: Recruiting | Type: Observational
Sponsor: University of Iowa (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH); Muscular Dystrophy Association (Other); University of Rochester (Other); University of Pennsylvania (Other); King's College Hospital NHS Trust (Other); Sydney Children's Hospitals Network (Other); Children's Hospital of Philadelphia (Other); University of Miami (Other); Johns Hopkins University (Other); Fondazione I.R.C.C.S. Istituto Neurologico Carlo Besta (Other); Cedars-Sinai Medical Center (Other); Nemours Children's Clinic (Other); Stanford University (Other); University of Minnesota (Other); Massachusetts General Hospital (Other); University of Colorado, Denver (Other); Children's National Research Institute (Other); University of Michigan (Other); St. Jude Children's Research Hospital (Other); Connecticut Children's Medical Center (Other); Seattle Children's Hospital (Other); The Hospital for Sick Children (Other)
Responsible Party: Principal Investigator, Michael Shy, Professor, University of Iowa
Other Study IDs: INC-6602; 1U54NS065712-01 (NIH)
Record Dates: First submitted 2010-08-09; First posted 2010-09-01 (Estimated); Last update posted 2025-10-07 (Actual); Status verified 2025-09

CONDITIONS: Charcot-Marie-Tooth Disease, Type Ia (Disorder); HMSN
Keywords: CMT; CMT1A
MeSH Terms: conditions — Charcot-Marie-Tooth Disease; Hereditary Sensory and Motor Neuropathy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — DNA extracted from whole blood. Filter cards with blood spots.
Oversight: Data Monitoring Committee: Yes | US Export: No

GROUPS / COHORTS (2):
- CMT1A: Families/people with genetically defined CMT1A
- Genetically undefined CMT: Families/people with genetically undefined CMT with common causes ruled out.

SUMMARY:
This project includes two projects. One is looking for new genes that cause Charcot Marie Tooth disease (CMT). The other is looking for genes that do not cause CMT, but may modify the symptoms a person has.

DETAILED DESCRIPTION:
This project is to understand modifier genes and how they influence the severity of disease expression, along with identifying new forms of CMT which have not been genetically determined. Subjects who are eligible will either have CMT type 1A (CMT1A) or an unknown form of CMT. Blood will be drawn and sent to the University of Miami where they receive the coded sample and process it through exome sequencing. Subjects will be told that this is optional.

ELIGIBILITY:
Inclusion Criteria:

All patients must agree to take part in the study and sign a consent form. A teenager (age 13-17 years) considering enrolling must agree to take part in the study and sign an assent form (depending on local ethics committee requirements).

Additional inclusion criteria are described below.

Inclusion Criteria: CMT1A Gene Modifier Study

Patients must have at least one of the following:

1. Patient has a documented PMP22 duplication. AND/OR
2. Patient has a first or second degree relative (parent, child, sibling, half- sibling, aunt, uncle, grandparent, grandchild, niece, or nephew) with a documented PMP22 duplication AND a clear link between that family member and the affected patient AND a phenotype consistent with CMT1A.

i. A clear link is necessary for a second-degree relative. For example, if a grandparent is affected and has a PMP22 duplication, and the parent does not have any signs, symptoms, or electrophysiology consistent with CMT1A, there is no clear link.

ii. In cases where clear links are not available, genetic testing is required for the patient or the first degree family member who is not clearly affected.

Inclusion Criteria - Patients for CMT Exome Project

a. Patient has demonstrated neuropathy on nerve conduction studies or clinically diagnosed genetic neuropathy, in the opinion of the investigator or genetic counsellor.

Inclusion Criteria - Controls for CMT Exome Project

1. Person is a family member of a CMT patient who is enrolled in the CMT Exome Project.

   AND one of the following:
2. Person does not have a peripheral neuropathy, in the opinion of the investigator or genetic counsellor.

   OR
3. Person is suspected to have a peripheral neuropathy, but has not been examined at an INC site.

Exclusion Criteria

1. Patient does not wish to participate or does not sign a consent form.
2. For CMT Exome Project, patient has a genetically confirmed form of CMT (i.e. mutation in MFN2 causing CMT2A, mutation in GARS causing CMT2D, etc.).
3. Patients with known neuropathy from a non-genetic source, such as chemotherapies (i.e. Vincristine, Taxol, Cisplatin), diabetes, alcoholism will be evaluated independently so that genetic contributions to their effects on CMT1A phenotypes can also be analyzed.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients participating in Inherited Neuropathies Consortium (INC)-6601 and meeting eligibility criteria for this study will be recruited.
Sampling Method: Non-Probability Sample
Enrollment: 1050 (Estimated)
Dates: Start 2010-05 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Charcot Marie Tooth disease type 1A (CMT1A) gene modifiers | once
  While the same genetic change - an extra copy of PMP22 - causes CMT1A by definition, it is unclear why some people have more severe symptoms and some have less severe. We are looking for genetic modifiers - changes in the DNA that may be causing the differences in symptoms.
New genetic causes of CMT | Once
  At least 33% of people with CMT have an unknown or genetically un-found form of the condition. We are looking for additional genes that cause CMT when mutated.

CONTACTS AND LOCATIONS:
Overall Officials: Michael E Shy, MD, Principal Investigator — University of Iowa
Locations (22):
- United States (17):
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Stanford University, Palo Alto, California
  - University of Colorado Hospital, Aurora, Colorado
  - Connecticut Children's Medical Center, Hartford, Connecticut
  - University of Miami, Miami, Florida
  - University of Iowa, Iowa City, Iowa
  - Johns Hopkins University, Baltimore, Maryland
  - Harvard/Massachusetts General Hospital, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - University of Minnesota, Maple Grove, Minnesota
  - University of Rochester, Rochester, New York
  - University of North Carolina, Chapel Hill, North Carolina
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - St. Jude Children's Research Hospital, Memphis, Tennessee
  - Houston Methodist Hospital, Houston, Texas
  - Seattle Children's Hospital, Seattle, Washington
- Children's Hospital of Westmead, Sydney, New South Wales, Australia
- The Hospital for Sick Children, Toronto, Ontario, Canada
- C. Besta Neurological Institute, Milan, Italy
- United Kingdom (2):
  - National Hospital of Neurology and Neurosurgery, London, England
  - Dubowitz Neuromuscular Centre, London

IPD SHARING:
Plan to Share IPD: Yes
De-identified RDCRN data is submitted to an ORDR-designated repository. For the current grant cycle, that repository has been dbGaP
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: (For Observational/Longitudinal/Natural History/Epidemiology studies): For the current grant cycle, available data will be released to the repository and will become available to the scientific community one year after publication of planned analyses, or after a period of 5 years from the date when the data were collected, whichever comes first.
Access Criteria: - For the current grant cycle, once de-identified data is posted on dbGaP, a summary of the study is posted and individual participant data is accessed via a request through dbGaP.
URL: https://www.ncbi.nlm.nih.gov/gap

REFERENCES:
- [Result] Montenegro G, Powell E, Huang J, Speziani F, Edwards YJ, Beecham G, Hulme W, Siskind C, Vance J, Shy M, Zuchner S. Exome sequencing allows for rapid gene identification in a Charcot-Marie-Tooth family. Ann Neurol. 2011 Mar;69(3):464-70. doi: 10.1002/ana.22235. Epub 2011 Jan 20. PMID 21254193
- See also: Inherited Neuropathies Consortium Website — https://www.rarediseasesnetwork.org/cms/inc